CLINICAL TRIAL: NCT04310436
Title: Modifying Unconscious Tongue Movements to Improve Fluency in Adults With a Confirmed Developmental Stammer. A Pilot Randomised Feasibility Study.
Brief Title: Modifying Unconscious Tongue Movements in Adults With Developmental Stammer.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher needing time off
Sponsor: Institute of Technology, Sligo (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITSligo HMcD
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Stammering
Keywords: Neuroplasticity; Eye saccades; Unconscious tongue movement
MeSH Terms: conditions — Stuttering | interventions — Air

STUDY DESIGN:
Intervention Model Description: Pilot Randomised Placebo Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Experimental Group instructed to modify saccadic origin by looking to naval for the start of the words dysfluencies were predicted
  Placebo Group instructed to modify saccadic origin by looking up for the start of the words dysfluencies were predicted
  Outcome assessor was blinded to treatment allocation. Participants Stammering behaviour to be assessed using SSI-4 a reliable validated objective measure of stuttering severity. Participants stammering behaviour is to be recorded via video link or in a separate lab and the assessor will be asked asked not to discuss the technique prescribed given to patients. Even if the patient mentioned the trials they would not discuss the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Looking down to naval. (Experimental): Modifying Saccade origin by looking down to naval.
  Interventions: Behavioral: Modifying saccades by looking down to naval.
- Looking up in the air. (Placebo Comparator): Modifying Saccade origin by looking up in the air.
  Interventions: Behavioral: Modifying saccades by looking in air.

INTERVENTIONS:
Behavioral: Modifying saccades by looking down to naval. — Paragraphs from list Provided by Researcher. Participants to read out loud for 10 minutes twice per day for the five week period. On any word they anticipate / experience dysfluencies look quickly down to their naval to reset the lateral tongue position.
  Arms: Looking down to naval.
Behavioral: Modifying saccades by looking in air. — Paragraphs from list provided by Researcher. Participants to read out loud for 10 minutes twice per day for the five week period. On any word they anticipate / experience dysfluencies look quickly up to reset the lateral tongue position.
  Arms: Looking up in the air.

SUMMARY:
This is a pilot randomised controlled trial investigating whether using modification of saccadic eye movements can control lateral unconscious tongue positioning and enhance fluency in adults with a confirmed developmental stammer. This study is being conducted as part of an MSc by research qualification at the Institute of Technology Sligo in Ireland with a view to extending to PhD. The setting is home setting with all assessments either taking place at home via video link or in the institute. The study is being conducted in conjunction with the Community Speech and Language Therapist and has attained ethical approval through Sligo University Hospital (SUH) Ethics Committee.

DETAILED DESCRIPTION:
Participants will be assessed for stammering severity either on line via video link or in the Institute of Technology Sligo Health Science & Exercise Physiology Lab (B2004) at three time points: before intervention, after a five-week trial period and three months post completion. Participants will complete two assessments at each time to cater for "off" days. Participants will be required to practice quick eye movements at the start of words / syllables where dysfluencies are predicted for 10 minutes twice a day for the treatment period. Training in eye movement (saccade) modification will occur following the initial assessment in IT Sligo, or video link.

Participants will be assigned to one of two treatment arms. An experimental arm, and a control (placebo) arm. All participants will be assessed regarding their premonitory awareness of anticipated dysfluencies both before training and at the three month Based on advice from Community Speech and language Manager (Ms Sinead Carthy), participants will voice/video message the principle investigator once per week for this five-week period to confirm compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adults age > 18 years.
* A diagnosis of confirmed developmental stammer from SALT characterized by stammering on ≥ 3% of syllables.
* A proficiency in the English Language.
* No diagnosis of any emotional, behavioural, learning or neurological disorder.
* Cognitive ability to take part.
* Have previously completed a course of outpatient treatment for confirmed developmental stammer.

Exclusion Criteria:

* Younger than 18 years.
* Not having completed a traditional intervention for stammer.
* This research is not intended to replace current interventions but provide additional possibilities for those adults who have completed a standard programme of intervention and their developmental stammer still persists and a rate of ≥ 3% of syllables

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Stammering Severity (SSI-4) (Howell et. al. 2011). | 10 minutes.
  Measures stuttering severity in adults and children. It measures the percentage of stuttered syllables versus fluent speech in the participant. It also measures the frequency of repetition and prolongations, duration of blocks, and physical concomitants.

SECONDARY OUTCOMES:
Stammering Experience Overall Assessment of the Speaker's Experience of Stuttering OASES-A (Yaruss & Quesal 2006). | 10 minutes.
  Measures the impact of stuttering on a person's life. Scores range between 1 (Mild) and 5 (Severe). The impact is broken down to four sections: General Information, Speaker's reactions, Daily Communication and Quality of life. There is also an overall impact score.
Premonitory Awareness in Stuttering Scale (PAiS) (Cholin et. al. 2016). | 10 minutes.
  Measures the anticipation effect in stuttering. 14 items assessing premonitory awareness of stuttering sensation to assess the individual's capacity, manner and style of anticipation. Each item consists of a 4-point Likert scale ranging from "not at all" to "very much". A higher score indicates a larger anticipation of stuttering by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Mc Donagh, MSc, Principal Investigator — Study Principal Investigator
Locations (1):
- Institute of Technology, Sligo, Sligo, Co Sligo, Ireland

DOCUMENTS (3):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT04310436/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT04310436/SAP_001.pdf
  • Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT04310436/ICF_002.pdf